CLINICAL TRIAL: NCT02681926
Title: VISITALY-Impact of a New Ablation Tracking Tool in Paroxysmal Atrial Fibrillation Ablation With Contact Force Technology
Brief Title: Impact of a New Ablation Tracking Tool in Paroxysmal Atrial Fibrillation Ablation With Contact Force Technology
Acronym: VISITALY
Status: Completed | Type: Observational
Sponsor: Giulio Zucchelli (Other)
Responsible Party: Sponsor-Investigator, Giulio Zucchelli, MD, PhD, Azienda Ospedaliero, Universitaria Pisana
Organization: Azienda Ospedaliero, Universitaria Pisana (Other)
Other Study IDs: 72607
Record Dates: First submitted 2016-02-03; First posted 2016-02-15 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2016-02

CONDITIONS: Catheter Ablation, Radiofrequency; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Average force group: A recent tool, called VISITAG, has been developed (and approved by EMEA) for Biosense Webster Navistar Smart Touch catheter in order to allow collection of ablation points with pre-determined characteristics, such as stability of catheter during ablation, mean contact force, drop in impedance. In the Average Force group, the operators decided to use the mean contact force as target parameter indicating a good lesion.
  Interventions: Procedure: VISITAG
- Force Time Integral group: In the Force Time Integral (FTI) group, the operators decided to use the FTI as target parameter indicating a good lesion.
  Interventions: Procedure: VISITAG

INTERVENTIONS:
Procedure: VISITAG — Paroxysmal atrial Fibrillation (PAF) ablation with contact force technology

SUMMARY:
Pulmonary vein isolation (PVI) is the cornerstone of atrial fibrillation (AF) ablation. A novel technology was recently developed to allow an automatic points annotation when indirect parameters of lesion formation reach predefined target values.

The aim of the study was to evaluate, in a prospective and multicenter study, the safety, efficiency and PVI effectiveness of a new ablation tracking tool (VISITAG; Biosense Webster) during paroxysmal AF ablation using a contact force sensing catheter.

DETAILED DESCRIPTION:
Background:

Catheter ablation is an effective treatment for paroxysmal atrial fibrillation (PAF) and pulmonary vein isolation is the most prevalent approach for catheter ablation of this kind of arrhythmia. Long-term success of the procedure is diminished by arrhythmia recurrences occurring predominantly because of reconnections in previously isolated pulmonary veins. The durability of pulmonary vein isolation is the cornerstone of the ablation and is influenced by transmurality and continuity of lesions. Limited animal and human studies suggest a correlation between electrode-tissue contact and radiofrequency lesion generation. Particularly, some contact forces (CFs) parameter (minimum contact force and minimum force time integral values) were strong predictors of gap formation in small studies . High contact force during ablation was also associated with the incidence of steam pop and with the subsequent risk of cardiac tamponade. A recent multicenter trial demonstrated that the irrigated CF-sensing catheter is safe and effective for the treatment of drug refractory symptomatic PAF, with no unanticipated device-related adverse events. The increased percent of time within investigator-targeted CF ranges correlated with increased freedom from arrhythmia recurrence. Stable CF during radiofrequency application increased the likelihood of 12-month success. Real-time measurement of contact force (CF) during catheter ablation of PAF has been recently confirmed to potentially impact procedural outcome, while in another small study, whatever CF visualization could assist operators in avoiding both low and high CF, CF-guided ablation did not affect AF recurrence. A recent tool, called VISITAG, has been developed (and approved by EMEA) for Biosense Webster Navistar Smart Touch catheter in order to allow collection of ablation points with pre-determined characteristics, such as stability of catheter during ablation, mean contact force, drop in impedance. The aim of this tool is to improve success rate of the procedure, reducing site of reconnections with a better understanding of lesion formation point by point, and in parallel to reduce complications, avoiding to give unnecessary ablation shots in sites already treated with a good set of lesions.

Purpose:

The aim of the study was to evaluate the effectiveness and safety of a strategy using a new ablation tracking tool (VISITAG; Biosense Webster) during PAF ablation with contact force technology.

Design:

Prospective, non-randomized, multicenter, registry

Medical Device:

Biosense Webster:

* Biosense Webster Smart Touch
* Biosense Webster CARTO3 (V3) system with VISITAG module.
* Biosense Webster CARTO3 system

Subject population:

Consecutive patients undergoing PAF ablation with abovementioned devices in several centers in Italy

Enrollment:

see in dedicated section

End-point:

see in dedicated section

Follow-up:

Follow-up will be performed using clinical visit with ECG, 12 hours ECG monitoring , loop recorder analysis or telephonic contact, following the centre strategy.

STATISTICAL ANALYSIS

Analysis Population:

All patients who are successfully registered will be included in the analysis.

Sample Size Calculations and Assumptions:

Being this an observational registry aiming at quantifying effect estimates without direct comparisons to literature benchmarks, the investigators relied on confidence interval profiling for sample size justification, without proceeding with formal power analysis. As the main analysis is a pooled analysis of patients with atrial fibrillation ablation, an overall and comprehensive analysis is planned as the primary analytical approach. Accordingly, the investigators computed that a target sample of 209 patients will enable the computation of reasonably precise 95% confidence intervals. Specifically, assuming a 12-month freedom from 72.5% AF/atrial flutter/atrial tachycardia recurrence at 1 year (in keeping with results of SMART-AF trial), confidence intervals computed with the adjusted Wald method would be 60% to 85% for a 209-patient sample (point estimate 151/209 [72.5%]).

Statistical Analysis:

Continuous endpoints will be summarized by presenting the total number of patients, mean, standard deviation, median, minimum, and maximum. Tabulation of categorical parameters will include counts and percentages. The outcomes will be summarized as both a discrete and a continuous variable using the method described above. Survival analysis (freedom from arrhythmia) will be performed with the Kaplan-Meier method. Statistical inference will be based on the computation of 95% confidence intervals using the adjusted Wald method. Additional analyses will involve key subgroups defined according to baseline, lesion, and procedural features, with statistical significance set at the 5% 2-tailed level. Specifically, Student t, Fisher exact, and log-rank tests will be used for such bivariate analyses, whereas multivariable linear regression, logistic regression, and Cox proportional hazard analyses will be used to adjust for confounders.

ELIGIBILITY:
Inclusion Criteria:

* PAF undergoing first ablation
* Patient was above the minimum age as required by local regulations to be participating in a registry regardless of gender and race;
* Provided Signed Informed Consent for the procedure.

Exclusion Criteria:

Patient had not to be included if any of the following conditions existed:

* Persistent or permanent atrial fibrillation;
* Redo ablation
* Age>75
* Left atrium diameter (LAD) > 50 mm
* Participation in another drug or device study that would have jeopardized the appropriate analysis of end-points of this study.
* High probability of non-adherence to the follow-up requirements (due to social, psychological or medical reasons)
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing PAF ablation with abovementioned devices in several centers in Italy
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-12; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation or other sustained atrial arrhythmias during 12 month after ablation, excluding 3 month of blanking period. | up to 12 months after ablation
  To determine the effectiveness at 12 month of a new ablation tracking tool called VISITAG (Biosense Webster) .
Freedom from major and minor complications during 1 month after ablation (SAFETY OUTCOME) | up to 1 month after ablation
  To determine the safety at 1 month of a new ablation tracking tool called VISITAG (Biosense Webster)

SECONDARY OUTCOMES:
Comparison of incidence of complications during 1 month after ablation using different VISITAG settings. | up to 1 month after ablation
  To assess safety of different VISITAG settings; to assess the role of visual gaps and VISITAG reaching preset target values in determining the safety
Freedom from atrial arrhythmias during 12 months after ablation (excluding 3 month blanking period) using different VISITAG settings. | up to12 months after ablation
  To assess the effectiveness of different VISITAG settings; to assess the role of visual gaps and VISITAG reaching preset target values in determining the effectiveness
Radiofrequency duration and procedural duration using different VISITAG settings. | procedure
  To assess efficiency of different VISITAG settings

CONTACTS AND LOCATIONS:
Locations (1):
- AOUPisana, Pisa, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided